CLINICAL TRIAL: NCT01889511
Title: Text Messaging to Improve Adherence to Oral Chemotherapy Agents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Yale University (Other); Sparrow Health System (Other); Diplomat Pharmacy (Unknown); Huron Medical Center (Other); Allegiance Health (Other); McLaren Cancer Institute (Unknown)
Responsible Party: Principal Investigator, Sandra Spoelstra, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R15CA176595 (NIH)
Record Dates: First submitted 2013-06-24; First posted 2013-06-28 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Cancer
Keywords: Text Messaging; Medication Adherence; Oral Agents
MeSH Terms: conditions — Neoplasms; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group - texts (Experimental): The intervention group will receive text messages for 21 days that are tailored to their oral agent regimen.
  Interventions: Behavioral: Intervention group - texts
- Control group (No Intervention): The control group will receive usual care, which consists of standard care and materials provided by the oncology office or pharmacy. In general, this includes instructions and information on the oral agent regimen (i.e., amount and timing), common side effects, how to manage symptoms, general ways to remember to take your pill (e.g., calendar or pill box), medication safety (i.e., storage), and how to contact a clinician for problems that arise.

INTERVENTIONS:
Behavioral: Intervention group - texts — Patients will be instructed to respond to the text message by sending a text stating if the oral agent was "taken". If there is no response after 15 minutes, a second text message will be sent out, again requesting a response. Satisfaction surveys will occur in the intervention group at week 5 when the text messages end; and will take five minutes.
  Arms: Intervention group - texts

SUMMARY:
The purpose of this Academic Research Enhancement Award proposal is to conduct a small-scale health-related research project on text messages to improve adherence to oral chemotherapy agents. Michigan State University College of Nursing has not been a major recipient of National Institute of Health grant funding. As a result, the overall objective of this proposal is to strengthen the research environment in the College of Nursing so that it can develop into a significant health-related scientific research enterprise. This project would involve undergraduate and graduate students, and thus, generate student interest in research as a career. The importance of the research planned for this proposal is as follows. More than 50 oral chemotherapy agents in pill form are currently on the market, with projections that in 3 years, 25% of cancer treatments will be delivered in pill form. For oral agents to achieve a therapeutically effective level for cancer treatment, patients must strictly adhere to the regimen. Adherence to oral cancer agents is often less than 80%, which may be inadequate for treating the cancer. To date, empirical research in the area of improving adherence to oral agents is underdeveloped. The goal of this research is to improve adherence to oral chemotherapy agents through a technology based strategy, tailored SMS text messages. This prospective randomized controlled trial will examine the feasibility, acceptability, and satisfaction with a 3-week tailored text message intervention for oral agent adherence. Descriptive statistics, generalized linear modeling, and generalized estimating equations will be used for analysis. In this proposal, preliminary data will be collected to examine efficacy of the text message intervention to promote adherence to oral agents. Data will then be used to further inform the development of an intervention to improve adherence to oral agents for an R01 application to conduct a larger randomized trial to test this innovative intervention. This study can have a transformative impact on oral agent adherence by developing a technology-based strategy to promote adherence among the increasing number of cancer patients who receive their cancer treatment in pill form. This type of novel intervention also has the potential to transform and impact many other ill populations that require adherence to a medication regimen.

DETAILED DESCRIPTION:
The therapeutic outcome of cancer treatment for patients taking oral chemotherapy agents depends heavily on adherence to the oral agent regimen. Yet recent research indicated that patients miss one-third of oral chemotherapy agent doses. With more than 50 oral anti-cancer agents on the market, it is projected that within 3 years, 25% of cancer treatment will be delivered in pill form. In this new treatment paradigm, care is moved from the clinics to home settings. This means that patients are seen less frequently by oncologists and greater responsibility is placed on the patients. Complicating this further, 75% of those with cancer also have comorbid conditions that require them to perform other self-care management (SCM) responsibilities. In addition, many have low self-efficacy, which may interfere with their ability to adhere to the oral agent. The therapeutic outcome for patients taking oral agents depends heavily on engaging patients to adhere to the regimen. Thus, a critical need exists to test novel interventions that promote adherence in patients taking oral chemotherapy agents.

The long-term goal of this research is to develop novel interventions to improve bio-behavioral outcomes of patients with cancer who have treatment in pill form. The objective of this study is to determine the feasibility, acceptability, satisfaction and efficacy of a short message service (SMS) text message intervention to promote adherence among cancer patients prescribed oral agents. The strategy to achieve this objective is to examine how technology can be used to improve adherence and to explore translation of these technologies to the clinical setting by deploying the following research plan.

This 10-week, 2-group, prospective randomized controlled trial will enroll 75 patients (50 in the intervention group and 25 in the control group), from 2 cancer centers, to test the feasibility and efficacy of a tailored intervention using text messages delivered to patient's cell phones to promote oral agent adherence. As these patients are newly prescribed an oral agent, they will be randomly assigned to either the intervention or the control group. At baseline (week 1), we will assess age, sex, race, cancer type and stage, self-efficacy, comorbid conditions and their SCM, and symptoms. For 21 days (week 2-4) the intervention group will receive a tailored text message for oral agent adherence plus usual care and the control group will receive only usual care. Each week (week 2-9) and at exit (week 10) an assessment of oral agent adherence and symptoms will occur. Satisfaction with the intervention will also be evaluated during the exit interview.

Specific Aims

Aim #1. To determine feasibility, defined as patient acceptance, retention in the study, and satisfaction, of a tailored text message intervention among patients who are on oral agents. Hypotheses to be tested are:

Hypothesis 1a: 80% of participants recruited will enroll in the study.

Hypothesis 1b: 80% of patients in the intervention group will complete 21 days of tailored text messages.

Hypothesis 1c: 90% of the intervention group will be satisfied with the tailored text messages.

Aim #2. To determine preliminary efficacy of the tailored text message intervention on adherence to oral agents. Hypotheses to be tested are:

Hypothesis 2a: The intervention group will have significantly higher rates of oral agent adherence than the control group.

Hypothesis 2b: There will be a large effect size of the intervention for group differences in adherence rates.

Exploratory aim: To explore the effect of oral agent complexity, low self-efficacy, symptom severity, comorbid conditions, and SCM of comorbid conditions on adherence to oral agents. We expect that adherence will be greater for patients with higher self-efficacy, simple oral agents, for those with fewer comorbid conditions, for those with fewer SCM responsibilities for their comorbid conditions, and for those with lower symptom severity.

This study can have a transformative impact on oral agent adherence by developing an easy-to-use, technology-based intervention to promote adherence among the increasing number of cancer patients whom receive treatment in this manner.

The significance of this study is that it targets a difficult clinical problem among patients who are very sick with a life threatening disease and must adhere to complex treatment protocols. This innovative intervention involves a readily available technology that can be used to interact with patients on a regular, consistent basis that would otherwise not be possible, feasible, or cost effective if done in a one-by-one interaction with a health care provider. The number of cancer patients who receive chemotherapy in pill form is increasing and this intervention will enable them to adhere and complete their cancer treatment. Thus, the intervention has high generalizability and the potential to transform care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer
* Prescribed an oncolytic or therapeutic oral agent (non-hormonal)
* Able to speak, read, and understand English
* Able and willing to receive phone calls
* Has a personal cell phone, and able and willing to receive and send a text message

Exclusion Criteria:

* Deaf, blind, or unable hear, or unable to accept phone calls
* Prescribed hormonal therapy for cancer treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility, defined as patient acceptance of a text message intervention among patients who are on oral agents. | Baseline to week-10.
  Feasibility of adherence to tailored text messages will be measured by the number of text messages delivered and any discontinuation of text messages during the course of the study while treatment with the oral agent is ongoing.
Feasibility, defined as retention in the study, among patients who are on oral agents. | Baseline.
  Acceptability of tailored text messaging will be measured by the number of patients who accept enrollment in the study compared to the number of patients who were offered to participate and by the percent of patients who complete the study. Acceptability will be assessed qualitatively by examining the reasons for attrition in the intervention group.
Feasibility defined as satisfaction with a text message intervention among patients who are on oral agents. | At week-4 after completion of text messages.
  Satisfaction with tailored text messages for adherence will be measured using a tool previously developed by this research team and administered in several previous studies that had Likert-scaled items. These Likert-scaled items will be modified for this study, adding items describing dimensions of satisfaction with the text messages. Satisfaction will be deemed high if the scores exceed 80%.

SECONDARY OUTCOMES:
Preliminary efficacy of the text message intervention on adherence to oral agents. | Calculated weekly from baseline to week 10; cumulative for the 10-week study period; and then intervention and control group are compared..
  Patients will be asked to recall and report the number pills taken (pill count) in the past 7 days at exit.
Preliminary efficacy of the text message intervention on adherence to oral agents. | Cumulative over the baseline to 10-weeks of the study then control and intervention groups are compared.
  The proportion of oral agent pills taken compared to what was prescribed will be calculated to determine the rate of adherence. Adherence will be examined at 3 levels: under-adherent (taking less than 85% of the prescribed dose); over-adherent (taking more than 100% of the prescribed dose in AM, PM, or both, or taking during rest periods); and adherent (taking between 85% and 100% of the medication); and cumulative.
Preliminary efficacy of the text message intervention on adherence to oral agents. | Cumulative over the baseline to 10-weeks of the study then control and intervention groups are compared..
  The relative dose intensity (RDI) will be calculated by examining the dose taken divided by standard dose intensity (prescribed number of pills) x 100.

OTHER OUTCOMES:
The effects of oral agent complexity, self-efficacy, symptom severity, and comorbid conditions on the intervention on adherence to oral agents. | Baseline and at 10 weeks in the study.
  The Cancer Self-Efficacy Scale (CASE), a self-report measure, will be administered (internal consistency reliability 0.95); Symptom Experience Inventory; and comorbidity presence on adherence as in stated measures

CONTACTS AND LOCATIONS:
Overall Officials: Sandra L Spoelstra, PhD, RN, Principal Investigator — Michigan State University
Locations (6):
- United States (6):
  - Yale University, New Haven, Connecticut
  - Diplomat Specialty Pharmacy, Flint, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Huron Medical Center, Port Huron, Michigan

REFERENCES:
- [Derived] Spoelstra SL, Given CW, Sikorskii A, Coursaris CK, Majumder A, DeKoekkoek T, Schueller M, Given BA. A randomized controlled trial of the feasibility and preliminary efficacy of a texting intervention on medication adherence in adults prescribed oral anti-cancer agents: study protocol. J Adv Nurs. 2015 Dec;71(12):2965-76. doi: 10.1111/jan.12714. Epub 2015 Jun 23. PMID 26100719